CLINICAL TRIAL: NCT03094403
Title: A Multi-Center, Double-Blind, Randomized, Placebo Controlled, Parallel-Group Study, Comparing Azeliac Acid Gel and Active Treatments to a Placebo Control in the Treatment of Moderate Facial Rosacea.
Brief Title: To Evaluate the Therapeutic Equivalence and Safety of Azelaic Acid 15% Topical Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AZAG 1533
Record Dates: First submitted 2017-03-17; First posted 2017-03-29 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — azelaic acid; Gels

STUDY DESIGN:
Intervention Model Description: Subjects in this randomized, double-blind, placebo controlled, parallel-group, multiple-center study will be randomly assigned in a 2:2:1 ratio to treatment with the test product, reference product or placebo control, respectively
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Azelaic Acid 15% topical gel (Experimental): Topical, twice daily, for 84 days A thin layer of study treatment was gently massaged into the affected areas on the face
  Interventions: Drug: Azelaic Acid 15% topical gel
- Finacea® (azelaic acid) Gel, 15% (Active Comparator): Topical, twice daily, for 84 days A thin layer of study treatment was gently massaged into the affected areas on the face
  Interventions: Drug: Finacea® (azelaic acid) Gel, 15%
- Placebo (Placebo Comparator): Topically to the face, twice a day A thin layer of study treatment was gently massaged into the affected areas on the face
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azelaic Acid 15% topical gel — Gel
  Other Names: Azelaic Acid
  Arms: Azelaic Acid 15% topical gel
Drug: Finacea® (azelaic acid) Gel, 15% — Gel
  Other Names: Azelaic Acid
  Arms: Finacea® (azelaic acid) Gel, 15%
Drug: Placebo — Gel
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
A Multi-Center, Double-Blind, Randomized, Placebo Controlled, Parallel-Group Study

DETAILED DESCRIPTION:
A Multi-Center, Double-Blind, Randomized, Placebo Controlled, Parallel-Group Study, comparing AZELAIC ACID TOPICAL GEL 15% TO FINACEA® and both active treatments to a Placebo Control in the treatment of Moderate of Facial Rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female ≥ 18 years-of-age with a clinical diagnosis of moderate facial rosacea;
* Subjects had to have a definite clinical diagnosis of facial rosacea severity Grade 3 as per the IGE

Exclusion Criteria:

* Female subjects who were pregnant, nursing, or planning to become pregnant during study participation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory lesion counts | 12 weeks
  Percent change from baseline to Week 12 in the inflammatory (papules and pustules) lesion counts

CONTACTS AND LOCATIONS:
Overall Officials: Catawba Research, Study Chair — http://catawbaresearch.com/contact/

IPD SHARING:
Plan to Share IPD: No